CLINICAL TRIAL: NCT01057979
Title: Motivational Interventions for Exercise in Hazardous Drinking College Students
Brief Title: Motivational Interventions for Lifestyle and Exercise in College Students
Acronym: MILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Linda Pescatello, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H09-043; R21AA017717-01A1 (NIH)
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Consumption
Keywords: exercise; college students; Sedentary college students
MeSH Terms: conditions — Alcohol Drinking; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MET + CM for Exercise (Experimental): Motivational Enhancement Therapy seeks to resolve ambivalence regarding exercise and increase intrinsic motivation to exercise. Contingency management offers tangible rewards for completing verified exercise.
  Interventions: Behavioral: MET + CM for Exercise
- MET + Exercise Contracting (Active Comparator): Motivational Enhancement Therapy seeks to resolve ambivalence regarding exercise and increase intrinsic motivation to exercise. Exercise contracting consists of weekly appointment to set specific goals for exercise in the upcoming week.
  Interventions: Behavioral: MET + Exercise Contracting

INTERVENTIONS:
Behavioral: MET + CM for Exercise — Motivational Enhancement Therapy seeks to resolve ambivalence regarding exercise and increase intrinsic motivation to exercise. Contingency management offers tangible rewards for completing verified exercise.
  Arms: MET + CM for Exercise
Behavioral: MET + Exercise Contracting — Motivational Enhancement Therapy seeks to resolve ambivalence regarding exercise and increase intrinsic motivation to exercise. Exercise contracting consists of weekly appointment to set specific goals for exercise in the upcoming week.
  Arms: MET + Exercise Contracting

SUMMARY:
Engagement in substance-free activities, such as exercise, has an inverse relationship to substance use in college students. While exercise has numerous physical and mental health benefits, the majority of college students are sedentary, infrequently engaging in exercise. Although exercise interventions to date often suffer from significant attrition and poor adherence, motivational interventions for exercise are beginning to show promise. In this pilot study we propose to develop and evaluate a novel exercise intervention combining Motivational Enhancement Therapy (MET) with contingency management (CM) in sedentary college students who use alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary college students who drink alcohol.

Exclusion Criteria:

* Medical contraindications for exercise.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Exercise engagement | 2 month, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah Weinstock, Ph.D., Principal Investigator — St. Louis University
Locations (1):
- University of Connecticut Storrs, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Weinstock J, Petry NM, Pescatello LS, Henderson CE. Sedentary college student drinkers can start exercising and reduce drinking after intervention. Psychol Addict Behav. 2016 Dec;30(8):791-801. doi: 10.1037/adb0000207. Epub 2016 Sep 26. PMID 27669095